CLINICAL TRIAL: NCT07115823
Title: A Longitudinal, Cohort Study Investigating the Impact of General Anaesthetic Caesarean Birth, With or Without ICU Admission, on Maternal Mental Health and Mother/Infant Bonding
Acronym: GABI
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Wellbeing of Women (Other); Burdett Trust for Nursing (Other)
Responsible Party: Sponsor
Other Study IDs: 359600; RTF1201 (Other Grant/Funding Number: Wellbeing of Women); RTF1201 (Other Grant/Funding Number: The Burdett Trust for Nursing)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: General Anaesthesia During Pregnancy
Keywords: General anaesthetic caesarean birth; Maternal mental health; Newborn bonding; Obstetric ICU admission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women or birthing people who have given birth by GACS: Women or birthing people aged 18 or older who have given birth by GACS in a UK hospital, within 12 months postpartum.
- Women or birthing people who have given birth by NACS: Women or birthing people aged 18 or older who have given birth by NACS in a UK hospital, within 12 months postpartum.

SUMMARY:
In the UK, approximately 6000 women every year undergo caesarean sections with general anaesthetic. Additionally, around 1300 women are admitted to Intensive Care Units (ICU) annually, typically due to pregnancy or childbirth complications. Some of these women are admitted to ICU for critical care immediately following a general anaesthetic caesarean section. However, there is little research on the impact of these experiences on women/birthing people and their families.

This project aims to explore the impact of general anaesthetic caesarean section, with or without subsequent ICU admission, on a mother's mental health and bonding with her newborn. Women and birthing people who have undergone a caesarean section with an epidural or spinal anaesthesia can also take part in this study, so that outcomes can be compared for different types of caesarean birth.

DETAILED DESCRIPTION:
Birth is a dynamic and transformative event, both on an individual and societal level and a key phase in the transition to motherhood. Many women or birthing people remain conscious during childbirth, allowing for immediate interaction and bonding activities with their newborns. However, those who undergo a General Anaesthetic Caesarean Section (GACS) are in a state of controlled unconsciousness due the effects of the general anaesthetic and therefore, will not experience their infant being born or early post-birth interactions.

Additionally, a small proportion of women or birthing people require admission to Intensive Care Units (ICU) following GACS. This can result in more prolonged periods where the mother is unable to emotionally connect or interact with her newborn. Consequently, this may increase the risk of mental health issues and affect bonding experiences for the mother postnatally. Yet, the impact of these events on women and their families remains largely underexplored.

This study Involves a longitudinal survey to collect prospective data on the experience of GACS compared to caesarean sections with neuraxial anaesthesia (NACS), focusing on mental health outcomes and maternal-infant bonding. The survey will include the Depression, Anxiety & Stress Scale (DASS-21), the City Birth Trauma Scale (CBTS) and the Postpartum Bonding Questionnaire (PBQ) and one question on self-harm from the Edinburgh Postnatal Depression Scale (EPDS). These measures will be collected upon completion of the initial survey and again 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over
* Gave birth by caesarean section (CS) in a UK hospital within the last 12 months
* Able and willing to access the internet
* ICU admission following CS

Exclusion Criteria:

* Under 18 years of age.
* Vaginal birth (including instrumental) that did not lead to GACS or NACS
* CS that has not taken place in a UK hospital
* CS more than 12 months ago
* ICU admission immediately following CS outside of the UK.
* Unable to access the internet

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any woman or birthing person who has undergone a caesarean section with general or neuraxial anaesthesia in a UK based hospital within 12 months postpartum.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Postnatal depression | 1-15 months post birth
  Depression scores (DASS-21)
Newborn bonding | 1-15 months post birth
  PBQ scores

SECONDARY OUTCOMES:
Anxiety | 1-15 months post birth
  Anxiety scores (DASS-21)
PTSD symptoms | 1-15 months post birth.
  City Birth Trauma Scale scores
Self-harm | 1-15 months post birth
  Scores from self-harm question on Edinburgh Postnatal Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Dr Hannah Rayment-Jones, Principal Investigator — King's College London
Locations (1):
- Faculty of Life Science and Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared as participants do not provide consent for the sharing of their data outside the research team, even in anonymised form.

REFERENCES:
- [Background] Wittkowski A, Vatter S, Muhinyi A, Garrett C, Henderson M. Measuring bonding or attachment in the parent-infant-relationship: A systematic review of parent-report assessment measures, their psychometric properties and clinical utility. Clin Psychol Rev. 2020 Dec;82:101906. doi: 10.1016/j.cpr.2020.101906. Epub 2020 Sep 3. PMID 32977111
- [Background] Wisner KL, Parry BL, Piontek CM. Clinical practice. Postpartum depression. N Engl J Med. 2002 Jul 18;347(3):194-9. doi: 10.1056/NEJMcp011542. No abstract available. PMID 12124409
- [Background] Widstrom AM, Brimdyr K, Svensson K, Cadwell K, Nissen E. Skin-to-skin contact the first hour after birth, underlying implications and clinical practice. Acta Paediatr. 2019 Jul;108(7):1192-1204. doi: 10.1111/apa.14754. Epub 2019 Mar 13. PMID 30762247
- [Background] Reck C, Hunt A, Fuchs T, Weiss R, Noon A, Moehler E, Downing G, Tronick EZ, Mundt C. Interactive regulation of affect in postpartum depressed mothers and their infants: an overview. Psychopathology. 2004 Nov-Dec;37(6):272-80. doi: 10.1159/000081983. Epub 2004 Nov 9. PMID 15539778
- [Background] Pownall M, Hutter RRC, Rockliffe L, Conner M. Memory and mood changes in pregnancy: a qualitative content analysis of women's first-hand accounts. J Reprod Infant Psychol. 2023 Nov;41(5):516-527. doi: 10.1080/02646838.2022.2052827. Epub 2022 Mar 20. PMID 35306947
- [Background] Powell DN, Leonhardt ND. A Longitudinal Examination of Mothers' Early Postnatal Adaptation: Relative Stability Across the First Eight Weeks. Matern Child Health J. 2023 Dec;27(12):2175-2184. doi: 10.1007/s10995-023-03776-4. Epub 2023 Sep 28. PMID 37768532
- [Background] NMPA Project Team. National maternity and perinatal audit: clinical report (2019) Based on births in NHS maternity services between 1st April 2016 and 31st March 2017. Royal College of Obstetrics and Gynaecology, London 2019. NMPA Clinical Report 2019.pdf (maternityaudit.org.uk)
- [Background] NMPA Project Team. National maternity and perinatal audit: clinical report (2021) Based on births in NHS maternity services between 1st April 2017 and 31st March 2018. Royal College of Obstetrics and Gynaecology, London 2019. NMPA Clinical Report 2019.pdf (maternityaudit.org.uk).
- [Background] Nakic Rados S, Matijas M, Kuhar L, Andelinovic M, Ayers S. Measuring and conceptualizing PTSD following childbirth: Validation of the City Birth Trauma Scale. Psychol Trauma. 2020 Feb;12(2):147-155. doi: 10.1037/tra0000501. Epub 2019 Aug 1. PMID 31368743
- [Background] National Maternity and Perinatal Audit Clinical Report 2022 Based on births in NHS maternity services in England and Wales between 1 April 2018 and 31 March 2019 Ref 336 NMPA Clinical Report_2022.pdf (maternityaudit.org.uk).
- [Background] Neczypor JL, Holley SL. Providing Evidence-Based Care During the Golden Hour. Nurs Womens Health. 2017 Dec;21(6):462-472. doi: 10.1016/j.nwh.2017.10.011. PMID 29223210
- [Background] Mehra R, Shebl FM, Cunningham SD, Magriples U, Barrette E, Herrera C, Kozhimannil KB, Ickovics JR. Area-level deprivation and preterm birth: results from a national, commercially-insured population. BMC Public Health. 2019 Feb 27;19(1):236. doi: 10.1186/s12889-019-6533-7. PMID 30813938
- [Background] Lovibond SH, Lovibond PF: Manual for the Depression Anxiety Stress Scales . 1995, Sydney , Psychology Foundation of Australia, 2nd.
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Krawczyk P, Jastrzebska A, Lipka D, Huras H. Pregnancy related and postpartum admissions to intensive care unit in the obstetric tertiary care center - an 8-year retrospective study. Ginekol Pol. 2021;92(8):575-578. doi: 10.5603/GP.a2021.0034. Epub 2021 Apr 12. PMID 33844261
- [Background] Knight M, B. K., Tuffnell D, Shakespeare J, Kotnis R, Kenyon S, Kurinczuk. (2022). Saving Lives, Improving Mother's Care Lessons learned to inform maternity care from the UK and Ireland Confidential Enquiries into Maternal Morbidity 2018-2020. Retrieved from https://www.npeu.ox.ac.uk/assets/downloads/mbrrace-uk/reports/maternal-report-2022/MBRRACE-UK_Maternal_MAIN_Report_2022_v10.pdf
- [Background] Handelzalts JE, Hairston IS, Matatyahu A. Construct Validity and Psychometric Properties of the Hebrew Version of the City Birth Trauma Scale. Front Psychol. 2018 Sep 18;9:1726. doi: 10.3389/fpsyg.2018.01726. eCollection 2018. PMID 30279671
- [Background] Grunberg VA, Geller PA, Hoffman C, Njoroge W, Ahmed A, Patterson CA. Parental mental health screening in the NICU: a psychosocial team initiative. J Perinatol. 2022 Mar;42(3):401-409. doi: 10.1038/s41372-021-01217-0. Epub 2021 Sep 27. PMID 34580422
- [Background] Ferguson S, Browne J, Taylor J, Davis D. Sense of coherence and women׳s birthing outcomes: A longitudinal survey. Midwifery. 2016 Mar;34:158-165. doi: 10.1016/j.midw.2015.11.017. Epub 2015 Dec 2. PMID 26689770
- [Background] Faulks F, Edvardsson K, Mogren I, Gray R, Copnell B, Shafiei T. Common mental disorders and perinatal outcomes in Victoria, Australia: A population-based retrospective cohort study. Women Birth. 2024 Mar;37(2):428-435. doi: 10.1016/j.wombi.2024.01.001. Epub 2024 Jan 12. PMID 38216393
- [Background] Farr SL, Dietz PM, O'Hara MW, Burley K, Ko JY. Postpartum anxiety and comorbid depression in a population-based sample of women. J Womens Health (Larchmt). 2014 Feb;23(2):120-8. doi: 10.1089/jwh.2013.4438. Epub 2013 Oct 26. PMID 24160774
- [Background] Edwards DR, Porter SA, Stein GS. A pilot study of postnatal depression following caesarean section using two retrospective self-rating instruments. J Psychosom Res. 1994 Feb;38(2):111-7. doi: 10.1016/0022-3999(94)90084-1. PMID 8189400
- [Background] De Schepper S, Vercauteren T, Tersago J, Jacquemyn Y, Raes F, Franck E. Post-Traumatic Stress Disorder after childbirth and the influence of maternity team care during labour and birth: A cohort study. Midwifery. 2016 Jan;32:87-92. doi: 10.1016/j.midw.2015.08.010. Epub 2015 Sep 8. PMID 26410818
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Chantry AA, Monnet C, Fresson J, Miller D, Bonnet MP, Deneux-Tharaux C. Repeated maternal ICU admission: Results from a nationwide analysis. Anaesth Crit Care Pain Med. 2021 Oct;40(5):100905. doi: 10.1016/j.accpm.2021.100905. Epub 2021 Jun 18. PMID 34153532
- [Background] Caparros-Gonzalez RA, Romero-Gonzalez B, Peralta-Ramirez MI, Ayers S, Galan-Paredes A, Caracuel-Romero A. Assessment of posttraumatic stress disorder among women after childbirth using the City Birth Trauma Scale in Spain. Psychol Trauma. 2021 Jul;13(5):545-554. doi: 10.1037/tra0001007. Epub 2021 Jan 28. PMID 33507792
- [Background] Brockington IF, Fraser C, Wilson D. The Postpartum Bonding Questionnaire: a validation. Arch Womens Ment Health. 2006 Sep;9(5):233-42. doi: 10.1007/s00737-006-0132-1. Epub 2006 May 4. PMID 16673041
- [Background] Brockington I. Postpartum psychiatric disorders. Lancet. 2004 Jan 24;363(9405):303-10. doi: 10.1016/S0140-6736(03)15390-1. PMID 14751705
- [Background] Roxanne B, Laura VDB, Yannic VG, Natacha VC, Luka VL, Kuipers YJ. Validation of the postpartum bonding questionnaire: A cross-sectional study among Flemish mothers. Midwifery. 2022 Apr;107:103280. doi: 10.1016/j.midw.2022.103280. Epub 2022 Feb 8. PMID 35182820
- [Background] Bhatia K, Columb M, Bewlay A, Eccles J, Hulgur M, Jayan N, Lie J, Verma D, Parikh R. The effect of COVID-19 on general anaesthesia rates for caesarean section. A cross-sectional analysis of six hospitals in the north-west of England. Anaesthesia. 2021 Mar;76(3):312-319. doi: 10.1111/anae.15313. Epub 2020 Nov 2. PMID 33073371
- [Background] Bell AF, Andersson E. The birth experience and women's postnatal depression: A systematic review. Midwifery. 2016 Aug;39:112-23. doi: 10.1016/j.midw.2016.04.014. Epub 2016 May 7. PMID 27321728
- [Background] Bamber JH, Lucas DN, Plaat F, Russell R. Obstetric anaesthetic practice in the UK: a descriptive analysis of the National Obstetric Anaesthetic Database 2009-14. Br J Anaesth. 2020 Oct;125(4):580-587. doi: 10.1016/j.bja.2020.06.053. Epub 2020 Jul 28. PMID 32736825
- [Background] Bamber JH, Goldacre R, Lucas DN, Quasim S, Knight M. A national cohort study to investigate the association between ethnicity and the provision of care in obstetric anaesthesia in England between 2011 and 2021. Anaesthesia. 2023 Jul;78(7):820-829. doi: 10.1111/anae.15987. Epub 2023 Mar 9. PMID 36893444
- [Background] Andersen LB, Melvaer LB, Videbech P, Lamont RF, Joergensen JS. Risk factors for developing post-traumatic stress disorder following childbirth: a systematic review. Acta Obstet Gynecol Scand. 2012 Nov;91(11):1261-72. doi: 10.1111/j.1600-0412.2012.01476.x. Epub 2012 Aug 13. PMID 22670573
- [Background] Ayers S, Wright DB, Thornton A. Development of a Measure of Postpartum PTSD: The City Birth Trauma Scale. Front Psychiatry. 2018 Sep 18;9:409. doi: 10.3389/fpsyt.2018.00409. eCollection 2018. PMID 30279664
- See also: NIHR South London Applied Research Collaboration — https://arc-sl.nihr.ac.uk/research-and-implementation/our-research-areas/maternity-and-perinatal-mental-health/exploring-1